CLINICAL TRIAL: NCT05074979
Title: Determining the Effectiveness of Telerehabilitation in COVID-19 Survivors
Brief Title: Telerehabilitation in COVID-19 Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Canan Demir, Research Assistant, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CDemir
Record Dates: First submitted 2021-10-03; First posted 2021-10-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COVID-19; Telerehabilitation
Keywords: COVID-19; telerehabilitation; COVID-19 Survivors; functional capacity; pulmonary functions; peripheral muscle oxygenation; home workout program
MeSH Terms: conditions — COVID-19 | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (Other): While other groups continue their exercise program for 6 weeks, this group will only be informed after COVID 19.
  Interventions: Other: informed program
- home exercise program group (Experimental): this group will implement COVID 19 home exercise program.
  Interventions: Other: home exercise program
- telerehabilitation group (Experimental): this group will implement COVID 19 telerehabilitation program.
  Interventions: Other: telerehabilitation

INTERVENTIONS:
Other: telerehabilitation — While telerehabilitation sessions will be applied to the participants in the telerehabilitation group for 6 weeks, home exercise program will be given to the home exercise program group and will be applied for 6 weeks.
  Arms: telerehabilitation group
Other: home exercise program — While telerehabilitation sessions will be applied to the participants in the telerehabilitation group for 6 weeks, home exercise program will be given to the home exercise program group and will be applied for 6 weeks.
  Arms: home exercise program group
Other: informed program — will informed after COVID 19
  Arms: control group

SUMMARY:
This study was carried out in the post-acute period of the telerehabilitation program in individuals with dyspnea who had COVID-19; It will be done to examine the effects on dyspnea, exercise capacity, respiratory functions, activities of daily living, muscle strength, muscle oxygenation, fatigue and quality of life parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COVID-19 by Computed Tomography (CT) or PCR test between the ages of 18-75,
* Do not have any orthopedic or neurological disease that will affect exercise capacity,
* Individuals who can take and execute verbal orders,
* Have had COVID-19 and at least 2 weeks have passed since the completion of the treatment,
* Individuals who have a computer or smart phone with a camera and internet connection and have the ability to use it (the participant himself or one of his family members living in the same house),
* Individuals who are sedentary (those whose physical activity level is inactive according to the Turkish version of the International Physical Activity Questionnaire (UFAA)),
* Having dyspnea at level 2 or 3 on the Medical Research Council Dyspnea Scale.

Exclusion Criteria:

* Those who have not had COVID-19 or acute period patients who are experiencing COVID-19,
* Individuals who cannot be contacted,
* Individuals with chronic heart disease,
* Those with concomitant uncontrolled disease; uncontrolled hypertension (resting blood pressure ≥160 /100mmHg), uncontrolled diabetes (random instantaneous blood glucose>16.7 mmol/l, HbA1C>7.0%),
* Those with concomitant severe organic disease (unstable hemodynamic heart disease, heart failure causing movement limitation, unstable angina, MI or other cardiac disease in the last 12 years),
* Individuals with cerebrovascular disease in the last 6 months,
* Those with digestive system ulcer, thyroid dysfunction or active stage of tuberculosis,
* Patients with Chronic Kidney Failure stage 3 and above according to Glomerular Filtration Rate (GFR),
* Individuals who have undergone intraraticular medication or surgery from their lower extremities in the last 6 months,
* Individuals who cannot walk independently,
* Individuals with any mental illness that may prevent them from living independently or receiving treatment,
* Uncooperative individuals for assessment and rehabilitation programs,
* Those with alcohol or substance addiction,
* Those who are pregnant, suspected of pregnancy or considering becoming pregnant,
* Participants in another study within the last 3 months or currently.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Severity of dyspnea assessment | 6 weeks
  Medical Research Council (MRC) Dyspnea Scale will be used to assess the severity of dyspnea. The severity of dyspnea during activities of daily living is graded from 0 to 4 on the Medical Research Council (MRC) Dyspnea Scale.
Physical activity level assessment | 6 weeks
  The physical activity level of the participants will be evaluated with the Turkish version of the "International Physical Activity Questionnaire" (UFAA).In the last 7 days with the survey; Vigorous physical activity (football, basketball, aerobics, cycling fast, lifting weights, carrying loads, etc.) time (min), Intermediate physical activity (light weight carrying, cycling at normal speed, folk dances, dancing, bowling, table tennis etc.) duration (min), walking and sitting times for one day (min) are questioned. All participants were given pre-study to assess the condition of being sedentary and those with inactive physical activity levels will be included in the study.
Cardiopulmonary endurance assessment | 6 weeks
  In order to evaluate cardiopulmonary endurance; A six-minute walking test will be applied. The test is 30 meters long, every 3 meters marked, the start and finish line are marked by a visible line, a smooth and straight done on the track. The distance the person walks for 6 minutes is recorded in meters.
Evaluation of peripheral muscle oxygenation | 6 weeks
  "Moxy muscle oxygen monitor" will be used to measure regional oxygen saturation (SmO2) and total hemoglobin (Thb) amount in capillaries under the muscle. Moxy muscle oxygen monitor (Fortiori Design LLC, USA) near infrared It is placed on the skin in a non-invasive way with spectroscopy (NIRS), It is a device that regional blood flow and measures oxygenation. A moxy muscle oxygen monitor will be attached to the quadriceps femoris muscle of the participants with a velcro and oxygenation measurements will be taken during both the dinelnim and 6-minute walking test.
Pulmonary function (slow vital capacity) | 6 weeks
  Single Breath Count Test will be used to evaluate slow vital capacity (the amount of air exhaled with slow exhalation after deep and maximal inspiration) and lung function. Single breath count (TNS), after maximal effort inhalation an individual with a metronome set to 2 beats per second in a normal speaking voice.
  It is a measure of how much you can count in your cadence.
Pulmonary function (Forced vital capacity (FVC)) | 6 weeks
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced vital capacity (FVC) will be evaluated.
Respiratory Muscle Strength | 6 weeks
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be measured using portable, electronic, oral pressure measuring device.
Activities of daily living assessment | 6 weeks
  Barthel Index will be used to evaluate activities of daily living.
Muscle strength assessment | 6 weeks
  Upper and lower extremity muscle strengths will be measured using a manual muscle strength measuring device.
Perceived fatigue assessment | 6 weeks
  Participants' perceived fatigue level will be recorded using the "Fatigue Scale". Developed by Borg, modified The category ratio scale (BORG CR-10 SCAL) with 10 degrees in shape is given to certain numbers.
  consists of corresponding definitions It will be recorded using the "Fatigue Scale". Developed by Borg, modified The category ratio scale (BORG CR-10 SCAL) with 10 degrees in shape is given to certain numbers consists of corresponding definitions. The Borg Scale is a subjective scale used to evaluate muscle fatigue.
General fatigue assessment | 6 weeks
  Participants will be asked to answer the chalder fatigue scale, which includes 11 questions about their fatigue in the past month. The maximum total score is 33; 4 and above scorers are described as tired.
Quality of life assessment | 6 weeks
  The Short Form-12 (SF-12) Questionnaire will be used to assess the quality of life.When scoring, two scores are obtained, the physical component and the mental component summary.
  is done. High scores indicate good health.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | 6 weeks
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced expiratory volume in the first second (FEV1) will be evaluated.
Pulmonary function (FEV1 / FVC) | 6 weeks
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, FEV1 / FVC will be evaluated.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%) | 6 weeks
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be evaluated.
Pulmonary function (Peak flow rate (PEF) | 6 weeks
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, peak flow rate (PEF) will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University, Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Balıkesir, Bandırma, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No